CLINICAL TRIAL: NCT07016646
Title: Combined Mental Health and Cash Transfer Intervention With Afghan Refugees in Turkiye
Brief Title: SH+ and Cash Assistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bogazici University (Other)
Responsible Party: Principal Investigator, Mitra Naseh, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202308168
Record Dates: First submitted 2025-04-04; First posted 2025-06-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stress; Depression Symptoms
Keywords: SH+; Cash Assistance; Afghan refugees; Turkiye
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled trial (RCT) will be conducted with a total of 40 participants. Participants will be randomly assigned to one of two groups: 20 individuals will receive both the Self-Help Plus (SH+) intervention and cash assistance, while the remaining 20 will receive cash assistance only and serve as the control group.
  One week after completing the intervention sessions, all participants-including those in the control group-will undergo post-intervention assessments, using the same questionnaires administered at baseline.
  To ensure ethical considerations and promote equity, the SH+ intervention will be offered to control group participants three months after the post-assessment.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded to their study arm due to the nature of the intervention, but outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: SH+ and cash assistance (Experimental): SH+: Self-Help Plus (SH+) is a five-session stress management program developed by the World Health Organization (WHO) for groups of up to 30 participants. It is facilitated by non-specialists who undergo brief training and use pre-recorded audio along with an illustrated guide, Doing What Matters in Times of Stress, to teach stress management techniques. Designed for adults experiencing stress, SH+ is adaptable to diverse living situations and circumstances. Research has demonstrated its effectiveness in alleviating psychological distress and preventing the onset of mental health disorders. Its flexible format makes it an excellent complement to other mental health interventions, whether as an initial step in a stepped care approach or as a community-based program integrated with broader community initiatives.
  Cash Assistance: A cash transfer of $300 or equal amount in Turkish Lira per participant ($60 or equal amount in Turkish Lira after each session)
  Interventions: Combination Product: Self-Help Plus (SH+) and cash transfer
- Control: Cash Assistance (Active Comparator): A cash transfer of $300 or equal amount in Turkish Lira per participant ($60 or equal amount in Turkish Lira each week for 5 weeks)
  Interventions: Other: Cash transfer

INTERVENTIONS:
Combination Product: Self-Help Plus (SH+) and cash transfer — SH+: Self-Help Plus (SH+) is a five-session stress management program developed by the World Health Organization (WHO) for groups of up to 30 participants. It is facilitated by non-specialists who undergo brief training and use pre-recorded audio along with an illustrated guide, Doing What Matters in Times of Stress, to teach stress management techniques. Designed for adults experiencing stress, SH+ is adaptable to diverse living situations and circumstances. Research has demonstrated its effectiveness in alleviating psychological distress and preventing the onset of mental health disorders. Its flexible format makes it an excellent complement to other mental health interventions, whether as an initial step in a stepped care approach or as a community-based program integrated with broader community initiatives.
  Cash Assistance: A cash transfer of $300 or equal amount in Turkish Lira per participant ($60 or equal amount in Turkish Lira after each session)
  Arms: Experimental: SH+ and cash assistance
Other: Cash transfer — A cash transfer of $300 or equal amount in Turkish Lira per participant ($60 or equal amount in Turkish Lira each week for 5 weeks)
  Arms: Control: Cash Assistance

SUMMARY:
This pilot project aims to evaluate the implementation outcomes and preliminary impacts of a combined low-intensity psychological intervention paired with cash assistance for Dari-speaking adult Afghan asylum-seeking women in Türkiye. The psychological intervention utilized is Self Help Plus (SH+), developed by the World Health Organization (WHO) for individuals in low-resource settings experiencing high stress levels.

This pilot, which builds on a previous needs assessment, will deliver the SH+ intervention through five two-hour sessions, supplemented by a cash transfer of USD 300 or equal amount in Turkish Lira per participant (USD 60 or equal amount in Turkish Lira after each session) to 40 Afghan asylum-seeking women in Türkiye.

The study will test the feasibility, acceptability, and practicality of the combined SH+ and cash transfer intervention and evaluate its effectiveness in addressing the mental health needs of forcibly displaced individuals through a two-arm randomized trial. The first group will receive SH+ and cash transfer simultaneously, and the second group will receive the cash transfer at the same time as the first group then receive the SH+ intervention after a 3-month delay.

Our local partners in Türkiye are the Afghan Refugees Solidarity Association (ARSA) and Boğaziçi University. We have already obtained IRB approval from Boğaziçi University.

DETAILED DESCRIPTION:
Afghan women asylum seekers and refugees who are already part of our ARSA's women's group will be screened for eligibility and enrollment in the study by a counselor from ARSA. The characteristics for recruited participants in this study will include a) being an Afghan refugee or asylum seeker residing in Türkiye, b) being a woman, c) being aged 18 or older, d) having the ability to read, speak, and consent in Dari, e) having high levels of psychological distress (scoring above 15 on the Kessler-10 Psychological Distress Scale [K-10]), and f) without an imminent risk of suicide (measured by the WHO PM+ assessment tool).

At the end of the screening questionnaire, eligible participants will receive a written consent form in both English and Dari. Qualified participants will also be provided with an informational presentation about the study and given a week to review the consent form carefully. Recruitment will continue until 40 eligible participants have provided consent.

Following the screening and consent process, 40 eligible participants will be randomized to two arms according to the 1:1 principle with automatized randomization software.

Group 1 (Receiving SH+ and cash transfer simultaneously):

Participants will complete the baseline assessment 1 week before the intervention. They will then participate in 5 weekly 2-hour SH+ session in person at ARSA in a private conference room. With each session, they will receive a $60 or equal amount in Turkish Lira in cash transfer. The program will be delivered by bilingual community facilitators who have completed a 3-day training on SH+ by WHO-certified SH+ trainers. Each session will follow the SH+ manual and the SH+ illustrated guide.

Childcare will be provided in a separate child-friendly room in ARSA during the sessions to remove barriers to participation and ensure that participants can participate in the sessions without concerns about their children's safety and well-being.

One week after the completion of the sessions, participants will complete the post-assessment, consisting of the same questionnaires used in the baseline assessment in addition to the measures related to implementation outcomes.

Group 2 (Receiving SH+ followed by cash transfer with a 3 month delay):

Participants will complete the baseline assessment 1 week before Group 1 begins their simultaneous intervention. While Group 1 is receiving their intervention, participants in Group 2 will receive a $60 or equal amount in Turkish Lira in cash transfer every week for 5 weeks. One week after the completion of Group 1's sessions, participants in Group 2 will complete the post-assessment, consisting of the same questionnaires used in the baseline assessment but without the implementation outcome measures.

After 3 months, participants in Group 2 will receive the SH+ intervention at ARSA (5 weeks, one 2-hour session per week, delivered by bilingual trained community facilitators, childcare provided at ARSA). One week after the completion of Group 2's sessions, participants in Group 2 will complete the full post-assessment, consisting of the same questionnaires used in the baseline assessment in addition to the measures related to implementation outcomes.

Supervision for facilitators will be provided by Zeynep Ilkkursun, a clinical psychologist in Türkiye. However, sessions will not be observed or recorded, and fidelity will be checked through conversations during the supervision sessions.

Additionally, semi-structured interviews will be conducted with the Afghan refugees who received the SH+ and the community members who were trained to deliver the intervention to get feedback on the content and clarity. Results will allow the study team to evaluate and understand the appropriateness and clarity of the procedures.

ELIGIBILITY:
Inclusion Criteria:

The characteristics for recruited participants in this study will include

1. being an Afghan refugee or asylum seeker residing in Türkiye,
2. being a woman,
3. being aged 18 or older,
4. having the ability to read, speak, and consent in Dari,
5. having high levels of psychological distress (scoring above 15 on the Farsi version of the Kessler-10 Psychological Distress Scale (K-10), and
6. without an imminent risk of suicide (measured by WHO PM+ assessment tool).

Exclusion Criteria:

* Having an imminent risk of suicide (measured by WHO PM+ assessment tool)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants identifying as adult female Afghan asylum seekers and refugees are eligible to participate
Enrollment: 40 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Kessler-10 Psychological Distress Scale (K-10) | Change from baseline (1 week before the intervention) to post assessment (6 weeks after the pre-assessment)
  Kessler-10 Psychological Distress Scale is a 10-item questionnaire that aims to measure psychological distress symptoms. Each of the 10 items are scored as 1, 2, 3, 4 and 5 to the response categories (1 = "none of the time" to 5= "all of the time"), providing a 10-50 severity score. Higher scores indicate higher levels of psychological distress. The Farsi version of the K-10 will be used in this study.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Change from baseline (1 week before the intervention) to post assessment (6 weeks after the pre-assessment
  Patient Health Questionnaire-9 is a 9 item questionnaire that aims to measure the severity of depression symptoms. Each of the 9 items are scored as 0, 1, 2, and 3 to the response categories (0 = "not at all," to 3= "nearly every day"), providing a 0-27 severity score. Higher scores indicate decreased functional status and increased symptom-related difficulties. The Farsi version of the PHQ-9 will be used in the study.
General Anxiety Disorder-7 (GAD-7) | Change from baseline (1 week before the intervention) to post assessment (6 weeks after the pre-assessment)
  General Anxiety Disorder-7 is a 7-item questionnaire that aims to measure anxiety symptoms. Each of the 7 items are scored as 0, 1, 2, and 3 to the response categories (0 = "not at all," to 3= "nearly every day"), providing a 0-21 severity score. Higher scores indicate higher levels of anxiety. The Farsi version of the GAD-7 will be used in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Afghan Refugees Solidarity Association ARSA, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No